CLINICAL TRIAL: NCT01073111
Title: Assessment of Neointimal Stent Strut Coverage and Endothelial Function After Second Generation Drug-Eluting Stent Systems
Brief Title: Assessment of Stent Strut Coverage and Endothelial Function After Drug-Eluting Stents
Acronym: ASSESS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Hyogo Medical University (Other)
Responsible Party: Principal Investigator, Kenichi Fujii, Assistant Professor, Hyogo Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASSESS
Record Dates: First submitted 2010-02-22; First posted 2010-02-23 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2017-02

CONDITIONS: Coronary Artery Disease; Atherosclerosis
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis

ARMS (3):
- zotarolimus-eluting stents (ENDEAVOR®) (Active Comparator)
  Interventions: Device: zotarolimus-eluting stent (ENDEAVOR®)
- sirolimus-eluting stents (CYPHER SELECT® PLUS) (Active Comparator)
  Interventions: Device: sirolimus-eluting stents (CYPHER SELECT® PLUS)
- everolimus-eluting stents (PROMUS®) (Active Comparator)
  Interventions: Device: everolimus-eluting stents (PROMUS®)

INTERVENTIONS:
Device: zotarolimus-eluting stent (ENDEAVOR®) — zotarolimus-eluting stent
  Arms: zotarolimus-eluting stents (ENDEAVOR®)
Device: sirolimus-eluting stents (CYPHER SELECT® PLUS) — sirolimus-eluting stents
  Arms: sirolimus-eluting stents (CYPHER SELECT® PLUS)
Device: everolimus-eluting stents (PROMUS®) — everolimus-eluting stents
  Arms: everolimus-eluting stents (PROMUS®)

SUMMARY:
The purpose of this study is to compare coronary endothelium function in patients with a zotarolimus-eluting versus a sirolimus-eluting or a everolimus-eluting stents with optical coherence tomography, vasoconstriction in response to acetylcholine, and coronary biomarker level.

ELIGIBILITY:
Inclusion Criteria:

* Significant coronary de novo lesion (> 70% by quantitative angiographic analysis)
* Patients with stable or acute coronary syndrome considered for coronary revascularization
* Reference vessel diameter of 2.5 to 3.5 mm by operator assessment

Exclusion Criteria:

* Contraindication to anti-platelet agents
* Ostial lesion within 5 mm from ostium
* Different DES in other vessel simultaneously
* Creatinine level 2.5 mg/dL
* Left main stenosis more than 50%.
* vein graft lesion
* Triple vessel disease with stenosis more than 50% in 3 epicardial coronary arteries
* Life expectancy 1 year
* Reference vessel < 2.5 mm or > 4.0 mm diameter by visual
* Long lesion that require more than three stents

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2011-10 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
To compare coronary endothelial function after primary angioplasty. | 6 months and 12 months
To compare the presence of neointimal stent strut coverage via optical coherence tomography. | 6 months and 12 months
To compare the serum biomarker levels measured in coronary artery blood. | 6 months and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hyogo College of Medicine, Nishinomiya, Japan